CLINICAL TRIAL: NCT02469792
Title: Effectiveness and Safety of Intraarticular Administration of Autologous Adipose-Derived Regenerative Cells for Treatment of Anterior Cruciate Ligament Partial Rupture
Brief Title: Effectiveness and Safety of Autologous ADRC for Treatment of Anterior Cruciate Ligament Partial Rupture
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Central Clinical Hospital w/Outpatient Health Center of Business Administration for the President of Russian Federation (Other Government)
Collaborators: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RU-CCH-03-01-14
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Anterior Cruciate Ligament Partial Rupture
Keywords: Anterior cruciate ligament; Ligament rupture; Intraarticular injection; ADRC; Adipose-derived regenerative cells; Adipose tissue; Stem cells
MeSH Terms: interventions — Lipectomy; Arthroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADRC injection (Experimental): Subjects will undergo liposuction under local anesthesia. Lipoaspirate will be processed to isolate and concentrate adipose-derived regenerative cells (ADRC). After ADRC isolation autologous cells suspension will be injected intraarticularly into anterior cruciated ligament.
  Interventions: Procedure: Liposuction; Device: ADRC isolation; Procedure: Arthroscopic surgery; Other: Intraarticular administration of autologous ADRC

INTERVENTIONS:
Procedure: Liposuction
Device: ADRC isolation — ADRC isolation performed using Celution 800/CRS System (Cytori Therapeutics Inc) according to manufacturer's protocol
Procedure: Arthroscopic surgery
Other: Intraarticular administration of autologous ADRC

SUMMARY:
Autologous adipose-derived regenerative cells (ADRC) will be extracted using Celution 800/CRS System (Cytori Therapeutics Inc) from a portion of the fat harvested from the patient's front abdominal wall. Patients will undergo knee arthroscopic surgery followed by one-time intraarticular ADRC administration (directly into anterior cruciate ligament). This is a single arm study with no control. All patients receive cell therapy.

DETAILED DESCRIPTION:
Patients with verified diagnosis partial rupture of anterior cruciate ligament will undergo liposuction from front abdominal wall under local anesthesia. After that autologous ADRC will be extracted using Celution 800/CRS System (Cytori Therapeutics Inc) from harvested adipose tissue. Same day patients will undergo knee arthroscopic surgery followed by one-time intraarticular freshly isolated ADRC administration (directly into anterior cruciate ligament close to the rupture).

ELIGIBILITY:
Inclusion Criteria:

* Patient suffers from partial rupture of anterior cruciate ligament (confirmed by MRI or knee arthroscopic surgery)
* Clinically significant knee instability (positive anterior drawer test, pivot shift test, and Lachman test)
* Patient is familiar with Participant information sheet
* Patient signed informed consent form

Non-inclusion Criteria:

* Knee osteoarthritis grade III and grade IV
* Medical history of autoimmune diseases
* Patients prescribed for immunosuppressive treatment
* Contraindications to the general or local anesthesia or medical history of allergic reactions to anesthetics
* Subcompensated or decompensated forms of chronic diseases of internal organs
* Significant weight loss (> 10% of body weight in the previous year) of unknown etiology
* Medical history of venous thromboembolism or estimated high risk of venous thromboembolism
* Clinically significant abnormalities in results of laboratory tests
* Any conditions limiting compliance (dementia, neuropsychiatric disease, drug and alcohol abuse etc.)
* Participation in other clinical trials (or administration of investigational drugs) during 3 months prior inclusion
* Patients with malignant tumors including postoperative period, patients receiving chemotherapy and/or radiotherapy.
* Patient's activated partial thromboplastin time exceeds normal levels more than 1,8 times
* Patients prescribed for anticoagulants treatment or patient received anticoagulants at least one hour prior lipoaspiration
* Medical history of heterotopic ossifications
* Patients prescribed for glycoprotein inhibitors treatment

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Patient's refusal from compliance with the requirements of contraception during the participation in research
* Chronic kidney disease IV - V stages (creatinine clearance < 30 mL/min estimated by Cockroft-Gault formula)
* Confirmed syphilis, HIV, hepatitis B or C infections

Dropout Criteria:

* Complete anterior cruciate ligament rupture confirmed by knee arthroscopic surgery
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Number of serious adverse events (SAEs) and serious adverse reactions (SARs) | 2 weeks after treatment

SECONDARY OUTCOMES:
Quality of life monitoring | Follow up to completion (up to 24 weeks after treatment)
  Quality of life estimated by validated questionnaires: the Short Form (36) Health Survey (SF-36), Knee Injury and Osteoarthritis Outcome Score (KOOS)
Knee pain intensity monitoring | Follow up to completion (up to 24 weeks after treatment)
  Knee pain intensity assessed by Visual Analogue Scale (no pain=0; maximum pain=100 mm)
Changes in knee joint structures | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee joint structure assessed by:
  1. X-ray (joint space width, bone contour, presence of osteophytes and sclerosis);
  2. MRI (articular cartilage, osteophytes, bone marrow abnormality, meniscal integrity, synovial effusion/tissue, anterior and posterior cruciate ligaments, and medial and lateral collateral ligaments);
  3. Ultrasonography (effusion, synovial thickening or hypertrophy, cartilage parameters, vascularity, Baker's cysts, osteophytes, tendon and ligament abnormalities, meniscal changes, bursitis, erosions and panniculitis)
Changes in knee function | Follow up to completion (up to 24 weeks after treatment)
  Changes in knee function assessed by questionnaire: Knee Society Score (KSS)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Ivannikov, Professor, Principal Investigator — I.M. Sechenov First Moscow State Medical University; Ilya I Eremin, MD, PhD, Principal Investigator — Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies
Locations (1):
- Federal State Budgetary Institution "Central Clinical Hospital with Outpatient Health Center" of the Business Administration for the President of the Russian Federation; Center for Biomedical Technologies, Moscow, Russia